CLINICAL TRIAL: NCT04778930
Title: Effectiveness of Physical Therapy for Improving the Functionality, Gait and Participation in the Environment in Children and Adolescents With Cerebral Palsy: Randomized Clinical Trial
Brief Title: Physical Therapy for Improving Functionality, Gait and Participation in Cerebral Palsy
Acronym: FIMAPACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Soraya Pacheco da Costa, University Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCosta
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Physical Therapy; Cerebral Palsy; Therapeutic Education; Telehealth
Keywords: Physical Therapy; Cerebral Palsy; Telehealth; Therapeutic Education
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities; Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As masking techniques, the persons responsible for the assessment of the subjects and the data collection, the random assignment and the intervention in each group will be independent from each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A_Intervention Group (Experimental): It will consist of 18 sessions, 3 times a week, for 6 consecutive weeks; on the one hand, 12 face-to-face sessions of approximately 90 minutes duration, in which the Physical Therapy treatment will be carried out based on training of specific tasks directed to objectives and training of gait with a treadmill; In addition, a therapeutic education program will be carried out, with 6 telehealth sessions lasting approximately 60 minutes, which will include action observation activities. The face-to-face sessions will be held at the Physical Therapy Teaching Unit at University of Alcalá, and the telehealth sessions of the Therapeutic Education program will be carried out by remote assistance through a digital platform. All will be carried out by specialist Physical Therapists, members of the research team.
  Interventions: Other: Physical Therapy; Other: THERAPEUTIC EDUCATION PROGRAM
- Group B_Control Group (Experimental): The subjects in this group will receive their usual Physical Therapy intervention regimen for 6 weeks at their referral center and the same telehealth Therapeutic Education program of the intervention group.
  Interventions: Other: THERAPEUTIC EDUCATION PROGRAM

INTERVENTIONS:
Other: Physical Therapy — FACE-TO FACE SESSIONS: approximately 90 minutes of Goal-directed training (activities for the activation of the muscles of the trunk, pelvis and lower limbs; and training of activities will be carried out in a functional and meaningful context, aimed at specific functional objectives, according to the interests of each participant and agreed with the participants and their families) and gait training on the treadmill for 20 minutes.
  TELEHEALTH THERAPEUTIC EDUCATION PROGRAM: Session 1: Concept and causes of CP, together with the general objectives and guidelines of the program. Session 2: The family-centered model; Sessions 3, 4 and 5: Actions Observation Therapy; Session 6: Program Evaluation.
  Other Names: Therapeutic Education; Family centered model; Action Observation Therapy; Goal-directed training; Treadmill
  Arms: Group A_Intervention Group
Other: THERAPEUTIC EDUCATION PROGRAM — TELEHEALTH THERAPEUTIC EDUCATION PROGRAM: Session 1: Concept and causes of CP, together with the general objectives and guidelines of the program. Session 2: The family-centered model; Sessions 3, 4 and 5: Actions Observation Therapy; Session 6: Program Evaluation.

SUMMARY:
Cerebral Palsy is a non-progressive nature lesion of the Central Nervous System, with a wide spectrum of impairments at body structure and function, which has a great impact at activity and participation in the environment. The intensity of participation is influenced by multiple factors, among which independent mobility stands out, through the functional activity of walking. Children and adolescents with Cerebral Palsy present limitations in gait function both at the level of body structure and activity and improving these aspects is one of the main therapeutic objectives in their treatment.

Physical Therapy interventions based on task learning and achieving objectives have proven to be effective in improving functional skills, gait and participation.

Due to COVID-19, interventions have been interrupted or reduced in periodicity. For this reason, it is essential to provide alternatives to Physical Therapy interventions for children and adolescents with Cerebral Palsy. Telehealth may play an important role both in maintaining function and in monitoring individuals, in addition to bringing the Physical Therapist closer to the natural environment of the child / adolescent through digital platforms.

Therefore the aim of this clinical trial is to verify that a Physiotherapy intervention that combines face-to-face sessions with telecare in natural settings is effective in improving the functional activity of walking and participation in the environment of children and adolescents with Cerebral Palsy.

The study population are children and adolescents diagnosed with Cerebral Palsy; ages 6-17 years old. The sample of 50 subjects (25 in each group) will be recruited in care centers for children and adolescents with Cerebral Palsy in Alcalá de Henares.

The outcome variables are: participation in the environment (Spanish version of the Children's Assessment of Participation and Enjoyment - CAPE), gait speed (10-meter walk test - 10MM), gait endurance (6-minute walk test - 6MM), gross motor function (Spanish version of the Gross Motor Function Measure - GMFM-SP) and static and dynamic balance (Spanish version of the Pediatric Balance Scale - PBS). They will be collected in three moments: baseline assessment (V0); intermediate assessment (V1) at 6 weeks at the end of each group intervention; Final assessment (V2) 3 months after baseline.

DETAILED DESCRIPTION:
Group A Physical Therapy intervention group will receive 18 sessions, 3 times a week, for 6 consecutive weeks; on the one hand, 12 face-to-face sessions of approximately 90 minutes duration, in which the Physical Therapy treatment will be carried out based on training of specific tasks directed to objectives and training of gait with a treadmill; In addition, a therapeutic education program will be carried out, with 6 telehealth sessions, which will include action observation therapy. Subjects in Group B (control group) will receive their usual Physiotherapy intervention regimen for 6 weeks at their referral center and the same telehealth Therapeutic Education program of the intervention group. The face-to-face sessions of the intervention group will be carried out in the Physiotherapy Teaching Unit of the University of Alcalá, and the telehealth sessions of the Therapeutic Education program of both groups will be carried out by remote assistance through a digital platform. All will be carried out by specialist Physiotherapists, members of the research team.

Statistical Analysis: After assessments, the data will be analyzed to verify the results. It will be done: descriptive analysis of the sample (means, medians, standard deviations and quartiles; normality test; frequency distributions): homogeneity check of the groups (t-Student or Mann Withney's U - quantitative variables; Chi square or F of Fisher - categorical variables); effectiveness analysis (parametric tests or not of paired samples; multivariate models to adjust for possible confounding factors; multivariate model of repeated measures to evaluate the result of the intervention. The statistical package Statistical Package for the Social Sciences software (25 version , SPSS Inc, Chicago, USA) or the statistical package STATA MP v14.2 (StataCo)

ELIGIBILITY:
Inclusion Criteria:

* GMFCS (I-III); MACS (I-III); CFCS (I-III)

Exclusion Criteria:

* having undergone surgery on lower limbs in the 6 months prior to his participation in the study; having surgery during the study; inability to follow the planned program due to moving to other city or other reason.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in baseline Environmental participation at 6 weeks and 3 months | Baseline assessment
  Spanish version of Children's Assessment of Participation and Enjoyment (CAPE)
Change in baseline Gait speed at 6 weeks and 3 months | Baseline assessment
  10 meter walk Test
Change in baseline Gait endurance at 6 weeks and 3 months | Baseline assessment
  6 minutes walk test
Change in baseline Gross Motor Function at 6 weeks and 3 months | Baseline assessment
  Spanish version of Gross Motor Function Measure (GMFM-SP)
Change in baseline Static and Dynamic Balance at 6 weeks and 3 months | Baseline assessment
  Spanish version of Pediatric Balance Scale (PBS)

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Pacheco da Costa, PhD, Principal Investigator — University Professor Physical Therapy Degree
Locations (1):
- Physiotherapy Neuromusculoskeletal in life stages Research Group - FINEMEV, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Result] Sellier E, McIntyre S, Smithers-Sheedy H, Platt MJ; SCPE and ACPR Groups. European and Australian Cerebral Palsy Surveillance Networks Working Together for Collaborative Research. Neuropediatrics. 2020 Apr;51(2):105-112. doi: 10.1055/s-0039-3402003. Epub 2020 Jan 7. PMID 31910452
- [Result] Schiariti V, Mahdi S, Bolte S. International Classification of Functioning, Disability and Health Core Sets for cerebral palsy, autism spectrum disorder, and attention-deficit-hyperactivity disorder. Dev Med Child Neurol. 2018 Sep;60(9):933-941. doi: 10.1111/dmcn.13922. Epub 2018 May 30. PMID 29845609
- [Result] Chakraborty S, Nandy A, Kesar TM. Gait deficits and dynamic stability in children and adolescents with cerebral palsy: A systematic review and meta-analysis. Clin Biomech (Bristol). 2020 Jan;71:11-23. doi: 10.1016/j.clinbiomech.2019.09.005. Epub 2019 Oct 18. PMID 31677546
- [Result] Toovey R, Bernie C, Harvey AR, McGinley JL, Spittle AJ. Task-specific gross motor skills training for ambulant school-aged children with cerebral palsy: a systematic review. BMJ Paediatr Open. 2017 Aug 11;1(1):e000078. doi: 10.1136/bmjpo-2017-000078. eCollection 2017. PMID 29637118
- [Result] Han YG, Yun CK. Effectiveness of treadmill training on gait function in children with cerebral palsy: meta-analysis. J Exerc Rehabil. 2020 Feb 26;16(1):10-19. doi: 10.12965/jer.1938748.374. eCollection 2020 Feb. PMID 32161730
- [Derived] Pacheco-da-Costa S, Rodriguez-Costa I, Abuin-Porras V, Asunsolo-Del-Barco A, Calvo-Fuente V, Soto-Vidal C. Effectiveness of Physiotherapy for Improving Participation, Gross Motor Function, Gait and Balance in Children and Adolescents with Cerebral Palsy: Study Protocol for a Randomized Controlled Trial. J Clin Med. 2025 Mar 24;14(7):2214. doi: 10.3390/jcm14072214. PMID 40217665